CLINICAL TRIAL: NCT02602249
Title: Phase 1 Study of Antigen-specific Cytotoxic T Lymphocytes Induced by Dendritic Cells Infected by Recombinant Adeno-associated Virus With MUC1 Gene(MUC1-gene-DC-CTL) or Directly Pulsed by MUC1 Peptide(MUC1-peptide-DC-CTL) in Gastric Cancer.
Brief Title: Clinical Safety and Preliminary Efficacy of MUC1-DC-CTL Treatment in Stage IV Gastric Cancer.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Doing Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Doing-003
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group A(control group) (No Intervention): saline infusion and follow up
- Experimental Group B (Experimental): MUC1-gene-DC-CTL will be used against tumor cells.
  Interventions: Biological: MUC1-gene-DC-CTL
- Experimental Group C (Experimental): MUC1-peptide-DC-CTL will be used against tumor cells.
  Interventions: Biological: MUC1-peptide-DC-CTL

INTERVENTIONS:
Biological: MUC1-gene-DC-CTL — MUC1-gene-DC-CTL will be used against tumor cells.
  Arms: Experimental Group B
Biological: MUC1-peptide-DC-CTL — MUC1-peptide-DC-CTL will be used against tumor cells.
  Arms: Experimental Group C

SUMMARY:
In this study, safety and effects of MUC1-gene-DC-CTL and MUC1-peptide-DC-CTL on human gastric cancer are going to be investigated.

DETAILED DESCRIPTION:
PBMC of the patient will be separated from peripheral blood.DCs infected by MUC1 and pulsed by MUC-1 peptide are made respectively from PBMC, then they are respectively cultured with T cells into MUC1-gene-DC-CTL and MUC1-peptide-DC-CTL which will be infused to the patients as immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male or female
* Age: from 18 to 80 years
* Histology: gastric cancer
* Clinical stage: stage IV
* Karnofsky performance status: more than 50%
* Expected survival: more than 2 months
* Laboratory tests results 7 days before the start of treatment:

  * White blood cells: more than 3.0 × 109/L
  * Platelets: more than 100 × 109/L
  * Neutrophils: more than 1.5 × 109/L
  * Hemoglobin: more than 80g/L
  * Serum glutamate pyruvate transaminase: less than 2.5 folds of the upper normal limit (ULN)
  * Serum glutamic-oxal (o) acetic transaminase: less than 2.5 × ULN
  * Serum bilirubin: less than 1.25 × ULN
  * Serum creatinine: less than 1.25 × ULN
* Pregnancy test: the test of women of child-bearing period must be negative 7 days before the start of treatment
* Contraception: male and female subjects of child-bearing period must adopt a reliable method of contraception before entry into this study until 30 days after stopping this study
* Informed consent: subject must have the ability to understand and voluntarily sign a written informed consent

Exclusion Criteria:

* History of neoplasms: other neoplasms
* Medical history: mental disease, or congestive heart failure, or severe coronary artery disease, or cardiac arrhythmias, or concomitant corticosteroid therapy
* Metastasis: clinical symptoms of brain metastasis
* Other clinical trial: the subject received other clinical trial before this study
* Laboratory tests: the serum test of human immunodeficiency virus, or hepatitis B virus, or hepatitis C virus was positive
* Woman: pregnant or lactating women
* Compliance: poor compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Reduced size of the tumor. | up to one year
  Tumor load will be evaluated by RECIST criteria.

SECONDARY OUTCOMES:
Safety, as measured by the rate of adverse events and serious adverse events | up to two years
  Safety, as measured by the rate of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: li gangyi, master, Study Chair — Beijing Doing Biomedical Co., Ltd.
Locations (3):
- China (3):
  - First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Huai'An First People'S Hospital, Huaian, Jiangsu
  - Beijing DOING Biomedical Co., Ltd, Beijing

IPD SHARING:
Plan to Share IPD: No